CLINICAL TRIAL: NCT03959917
Title: Bipolar Transurethral Resection of the Prostate; Complications and Possibility to do as Outpatient Procedure
Brief Title: TURP; Complications and Outpatient Care
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Other Study IDs: EPN 201801-12
Record Dates: First submitted 2019-05-21; First posted 2019-05-22 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: prostate; resection; incontinence; erectile dysfunction
MeSH Terms: conditions — Prostatic Hyperplasia; Erectile Dysfunction | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: transurethral resection of the prostate — Surgical removal of benign prostatic tissue
  Other Names: TUR P

SUMMARY:
This study aims to investigate the impact of transurethral prostate resection in regard to complications. These are direct surgical complications, such as bleeding, infection and readmissions, as well as the long term complications as incontinence and impotence. Also, the study aims to investigate if selected cases of patients could be performed as outpatient surgery, thereby reducing cost.

DETAILED DESCRIPTION:
Transuretral prostate resection (TUR P) is a common procedure to relieve voiding problems in men. After the introduction of bipolar resection with saline, the serious complication of transurethral resection syndrome (i.e. acute hypo-natremia) has been eradicated.

The post surgical care is generally a couple of days inhospital care. The reson for this, is the risk of clot formation and in rare cases post surgical infection.

However, in selected cases, outpatient surgery has been performed with encouraging results. However, the technique has not been spread widely. The use of ambulatory surgery would reduce the direct cost of the procedure, thereby increasing it´s availability.

Also, complications in contemporary TUR P in the modern era (outside of the selected patients of clinical trials) is lacking. The information of complications that can be expected is therefore an important for patient counseling. In some studies, the use of incontinence pads after TUR P is more than 15%, which is important to reliably ascertain if this is holds true.

ELIGIBILITY:
Inclusion Criteria:

* Planned for transurethral resection of the prostate (TUR P)

Exclusion Criteria:

* No consent to participate

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a feasibility cohort study. All patients planned for TUR P are eligible. Patients in the ambulatory group have prostate size less than 50 cc and ASA score less less than 4 and ser under 80 years of age. This is clinical routine at the study site.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-05-15 (Estimated); Primary Completion 2020-02-15 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients able to be discharged the day of surgery | One day
Proportion of patients readmitted to hospital the first day of surgery | One day

SECONDARY OUTCOMES:
Change in IPSS score | 6 months
  International prostate symptom score, range 0-35
Number of patients with cancer in surgical specimen | 6 months
  Pathological confirmed prostate cancer, all Gleasson Grades (6-10)
Readmission rates within 30 days of surgery | 30 days
Complications | 30 days
  Clavien Dindo Classification
Proportion catheter free | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Östersunds hospital, Östersund, Jämtland County, Sweden